CLINICAL TRIAL: NCT01223859
Title: The Impact of Pretreatment Assessment of Oropharynx on Interstitial Soft Palate Radiofrequency Surgery Outcome - a Multi-center Study in Patients With Habitual Snoring
Brief Title: Pretreatment Assessment of Oropharynx Ans Soft Palate Radiofrequency Surgery - a Multi-center Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Olympus Surgical Technologies Europe, Celon Ag Medical Instruments, Teltow, Germany (Unknown); Helsinki University Central Hospital (Other)
Responsible Party: Leif Bäck MD, PhD, Dept of ORL HN Surgery
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: lefa
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2007-10

CONDITIONS: Snoring
Keywords: Radiofrequency, ablation, RFA, RFTA, RFITT, soft palate.
MeSH Terms: conditions — Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intervention (Experimental): Interstitial soft palate RF surgery
  Interventions: Procedure: Interstitial soft palate surgery

INTERVENTIONS:
Procedure: Interstitial soft palate surgery — Soft palate RF surgery in local anaesthesia
  Other Names: RFA; RFTA

SUMMARY:
Interstitial radiofrequency (RF) surgery of the soft palate (SP) is an established option in the treatment of habitual snoring. The decision making process in the management of habitual snoring would benefit from diagnostic guidelines for oropharyngeal findings. The aim was to investigate the correlation of systematic clinical pretreatment oropharyngeal examination scores with the efficacy of interstitial RF surgery of SP in a multi-center study

DETAILED DESCRIPTION:
TABLE 1. The inclusion and exclusion criterion used for the multicenter study.

Criteria Inclusion Exclusion _____________

Age (years) 18-65 < 18, > 65

Habitual snoring yes no Excessive daytime sleepiness no yes

BMI (kg/m2) < 28 > 28

AHI (events/hour) < 15 > 15

Overjet (mm) < 5 > 5 Clinical suspicion of obstruction no yes at base of tongue

Size of palatine tonsils (grade) 0-II III-IV

Nose breathing problems no yes

Pharyngeal tonsil hypertrophy no yes

A bed partner to assess snoring yes no

_____________

Abbreviations: BMI = body mass index, AHI = apnea-hypopnea index.

ELIGIBILITY:
TABLE 1. The inclusion and exclusion criterion used for the multicenter study.

Criteria Inclusion Exclusion _____________

Age (years) 18-65 < 18, > 65

Habitual snoring yes no Excessive daytime sleepiness no yes

BMI (kg/m2) < 28 > 28

AHI (events/hour) < 15 > 15

Overjet (mm) < 5 > 5 Clinical suspicion of obstruction no yes at base of tongue

Size of palatine tonsils (grade) 0-II III-IV

Nose breathing problems no yes

Pharyngeal tonsil hypertrophy no yes

A bed partner to assess snoring yes no

_____________

Abbreviations: BMI = body mass index, AHI = apnea-hypopnea index.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2008-01; Primary Completion 2009-07 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
VAS | 3 months postoperatively
  Visual analogue scale snoring patient and bed partner

CONTACTS AND LOCATIONS:
Overall Officials: Leif JJ Bäck, MD PhD, Study Director — Helsinki University Dept of ORL HN Surg

REFERENCES:
- [Derived] Back LJ, Koivunen P, Pyykko I, Stene BK, Makitie AA. The impact of pretreatment assessment of oropharynx on interstitial soft palate radiofrequency surgery outcome--a multi-center study in patients with habitual snoring. Sleep Breath. 2012 Mar;16(1):199-204. doi: 10.1007/s11325-011-0490-4. Epub 2011 Feb 12. PMID 21311985